CLINICAL TRIAL: NCT00956319
Title: A Randomized, Open-Label, Active-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Zolpidem Modified Release (MR) in Patients With Primary Insomnia
Brief Title: A Study to Evaluate Efficacy and Safety of Zolpidem Modified Release Formulation in Insomnia Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STCR-0802-TW
Record Dates: First submitted 2009-08-09; First posted 2009-08-11 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Sleep Initiation and Maintenance Disorders; Primary Insomnia
Keywords: Insomnia; Zolpidem; Estazolam
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Estazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zolpidem group (Experimental)
  Interventions: Drug: Zolpidem MR
- Estazolam group (Active Comparator)
  Interventions: Drug: Estazolam

INTERVENTIONS:
Drug: Zolpidem MR — oral
  Other Names: Stilnox CR; Ambient CR
  Arms: Zolpidem group
Drug: Estazolam — oral
  Other Names: Eurodin
  Arms: Estazolam group

SUMMARY:
The purpose of the study is to investigate the efficacy and safety of zolpidem modified release (MR) tablet using estazolam (Eurodin) as a comparative drug in patients with primary insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary insomnia based on DSM-IV criteria (307.42)
* Written informed consent has been obtained

Exclusion Criteria:

* Patients with sleep apnea syndrome, narcolepsy, presence or suspicion of periodic leg movement or restless leg syndrome
* Patients with hepatic failure, myasthenia gravis, or hypersensitivity to zolpidem
* Patients who are known to be current drug or alcohol abuser or likely to concomitantly consume alcoholic beverages (more than 3 times/week)
* Patients who are pregnant, lactating or intend to become pregnant during the study period
* Patients who have received antidepressants or anxiolytics will not allow to change the dose or discontinue the previous medication throughout the study
* Any clinically significant condition, which in the opinion of the investigator makes the patients unsuitable for the trial
* Participation in any clinical trial within 1 month prior to randomization

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2009-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Total score of Pittsburgh Sleep Quality Index (PSQ) | 3 weeks

SECONDARY OUTCOMES:
Physician's clinical global impression (CGI) | 3 weeks
Patient's global impression (PG) | 3 weeks
Sleep latency, total sleep time, number of awakenings, wake time after sleep onset as derived from sleep diary | 3 weeks
Incidence and severity of adverse events, including abnormal sleep behavior | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Taipei, Taiwan